CLINICAL TRIAL: NCT03478956
Title: A Phase I, Open-Label, Randomized, Pharmacokinetic, Pharmacodynamic, and Safety Study of Etrolizumab Followed by Open-Label Extension and Safety Monitoring in Pediatric Patients From 4 Years to Less Than 18 Years Of Age With Moderate to Severe Ulcerative Colitis or Moderate To Severe Crohn's Disease
Brief Title: A Phase I Study of Etrolizumab Followed by Open-Label Extension and Safety Monitoring in Pediatric Patients With Moderate to Severe Ulcerative Colitis or Moderate to Severe Crohn's Disease
Acronym: FENNEL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to program discontinuation, based on mixed efficacy results in the adult ulcerative colitis and Crohn's disease studies. There were no safety concerns.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA40192; 2017-003649-10 (EudraCT Number)
Record Dates: First submitted 2018-03-26; First posted 2018-03-27 (Actual); Results first posted 2020-08-05 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — etrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etrolizumab Q4W (Experimental): Etrolizumab 1.5 milligrams per kilogram of body weight (mg/kg) was administered by subcutaneous (SC) injection once every 4 weeks (Q4W) for a total of 4 doses over the course of the 24-week randomized treatment phase (16-week treatment period plus 8-week safety follow-up). Participants were then given the option to participate in the 312-week open-label extension (OLE) treatment phase with etrolizumab 1.5 mg/kg SC Q4W followed by the 104-week safety surveillance phase (no etrolizumab treatment) to monitor for progressive multifocal leukoencephalopathy (PML). All participants who chose not to enter the OLE phase after the 24-week randomized treatment phase entered the 104-week PML monitoring phase.
  Interventions: Drug: Etrolizumab
- Etrolizumab Q8W (Experimental): Etrolizumab 3.0 mg/kg was administered by subcutaneous (SC) injection once every 8 weeks (Q8W) for a total of 2 doses over the course of the 24-week randomized treatment phase (16-week treatment period plus 8-week safety follow-up). Participants were then given the option to participate in the 312-week open-label extension (OLE) treatment phase with etrolizumab 1.5 mg/kg SC Q4W followed by the 104-week safety surveillance phase (no etrolizumab treatment) to monitor for progressive multifocal leukoencephalopathy (PML). All participants who chose not to enter the OLE phase after the 24-week randomized treatment phase entered the 104-week PML monitoring phase.
  Interventions: Drug: Etrolizumab

INTERVENTIONS:
Drug: Etrolizumab — Etrolizumab was administered by subcutaneous (SC) injection as described for each treatment arm.
  Other Names: RG7413; RO5490261; PRO145223; rhuMAb Beta7

SUMMARY:
This study will evaluate pharmacokinetics, pharmacodynamics and safety of etrolizumab in pediatric patients of 4 to <18 years of age with moderate to severe ulcerative colitis (UC) or with moderate to severe Crohn's disease (CD).

ELIGIBILITY:
Inclusion Criteria:

* Age of 4 years to <18 years at the time of signing the Informed Consent Form.
* Weight of 13 kilograms (kg) or more
* Diagnosis of ulcerative colitis (UC) or Crohn's Disease (CD) confirmed by biopsy and established for ≥3 months (i.e., after first diagnosis by a physician according to American College of Gastroenterology [ACG] guidelines) prior to screening
* Inadequate response, loss of response or intolerance to prior immunosuppressants and/or corticosteroid treatment and/or anti-tumor necrosis factor (TNF) therapy
* For postpubertal females of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive methods during the treatment period and for at least 24 weeks after the last dose of etrolizumab.
* For male patients: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

* Pregnant or lactating
* Lack of peripheral venous access
* Congenital or acquired immune deficiency
* Neurological conditions or diseases that may interfere with monitoring for progressive multifocal leukoencephalopathy (PML)
* History of demyelinating disease
* History of cancer, including hematologic malignancy, solid tumors, and carcinoma in situ, within 5 years before screening

Exclusion Criteria Related to Inflammatory Bowel Disease:

* Prior extensive colonic resection, subtotal or total colectomy, or planned surgery
* Past or present ileostomy or colostomy
* Diagnosis of indeterminate colitis
* Suspicion of ischemic colitis, radiation colitis, or microscopic colitis
* Diagnosis of toxic megacolon within 12 months of initial screening visit
* Abdominal abscess
* A history or current evidence of colonic mucosal dysplasia
* Patients with fixed symptomatic stenosis of the intestine
* Patients with history or evidence of adenomatous colonic polyps that have not been removed

Exclusion Criteria Related to Ulcerative Colitis:

* Severe extensive colitis per investigator judgment that colectomy is imminent

Exclusion Criteria Related to Crohn's Disease:

* Sinus tract with evidence for infection (e.g., purulent discharge) in the clinical judgment of the investigator
* Short-bowel syndrome
* Evidence of abdominal or perianal abscess
* Expected to require surgery to manage CD-related complications during the study

Exclusion Criteria Related to Prior or Concomitant Therapy:

* Any prior treatment with anti-integrin agents (including natalizumab, vedolizumab, and efalizumab), ustekinumab, anti-adhesion molecules (e.g., anti-MAdCAM-1), or rituximab
* Use of IV steroids within 30 days prior to screening with the exception of a single administration of IV steroid
* Use of agents that deplete B or T cells (e.g., alemtuzumab or visilizumab) within 12 months prior to Day 1, with the exception of AZA and 6-MP
* Use of cyclosporine, tacrolimus, sirolimus, or mycophenolate mofetil (MMF) within 4 weeks prior to Day 1
* Use of other biologics (e.g. anti-TNF) within 8 weeks before dosing (unless drug level is below detectability before completion of the 8-week interval)
* Chronic nonsteroidal anti-inflammatory drug (NSAID) use
* Patients who are currently using anticoagulants
* Apheresis (i.e., Adacolumn apheresis) within 2 weeks prior to Day 1
* Received any investigational treatment including investigational vaccines within 12 weeks prior to Day 1 of the study or 5 half-lives of the investigational product, whichever is greater
* History of moderate or severe allergic or anaphylactic/anaphylactoid reactions to chimeric, human, or humanized antibodies, fusion proteins, or murine proteins or hypersensitivity to etrolizumab (active drug substance) or any of the excipients (L-histidine, L-arginine, succinic acid, polysorbate 20)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Hôpital Enfants Reine Fabiola, Brussels, Belgium
- Poland (2):
  - Gabinet Lekarski, Bartosz Korczowski, Rzeszów
  - Centrum Zdrowia MDM, Warsaw
- Hospital Niño Jesus; Servicio de Pediatria - Gastrenterologia y Nutricion, Madrid, Spain
- Royal Manchester Childrens Hospital, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in 3 parts: Randomized Treatment Period, Open-label Extension (OLE) Period and Progressive Multifocal Leukoencephalopathy (PML) Safety Monitoring (SM) Period. Participants who completed the randomized treatment period were given the option to continue treatment in OLE period. After the randomized treatment period (if they did not enter OLE) or after the OLE period, participants were given the option to continue in PML SM period during which they were monitored for PML.
Groups:
- Etrolizumab Q4W: Etrolizumab 1.5 milligrams per kilogram of body weight (mg/kg) was administered by subcutaneous (SC) injection once every 4 weeks (Q4W) for a total of 4 doses over the course of the 24-week randomized treatment phase (16-week treatment plus 8-week safety follow-up).
- Etrolizumab Q8W: Etrolizumab 3.0 milligrams per kilogram of body weight (mg/kg) was administered by SC injection once every 8 weeks (Q8W) for a total of 2 doses over the course of the 24-week randomized treatment phase (16-week treatment plus 8-week safety follow-up).
- OLE: Etrolizumab 1.5 mg Q4W: Participants from Etrolizumab Q4W and Etrolizumab Q8W who completed the randomized treatment period, were given the option to participate in the OLE period. All participants who chose to enter the OLE period were administered etrolizumab 1.5 mg/kg SC Q4W for a maximum of 183 weeks. Post treatment discontinuation participants entered a 12-week safety follow up.
- PML Safety Monitoring: After the randomized treatment period (if participants did not enter the OLE period) or after the OLE period, participants who chose to continue in PML safety surveillance phase were monitored for PML for approximately 92 weeks. Participants who chose to enter PML surveillance phase were only followed up for PML and did not receive any study treatment.
Period: Randomized Treatment Period
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W | OLE: Etrolizumab 1.5 mg Q4W | PML Safety Monitoring
Started (Enrolled in Randomized Treatment Phase) | 12 | 12 | 0 | 0
Received at Least One Dose of Study Drug | 12 | 12 | 0 | 0
Completed Treatment | 11 | 10 | 0 | 0
Completed | 11 | 11 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Open Label Extension Period
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W | OLE: Etrolizumab 1.5 mg Q4W | PML Safety Monitoring
Started | 0 | 0 | 21 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 21 | 0
Not completed — Adverse Event | 0 | 0 | 4 | 0
Not completed — Lack of Efficacy | 0 | 0 | 8 | 0
Not completed — Reason Not Provided | 0 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 6 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0
Period: PML Safety Monitoring Period
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W | OLE: Etrolizumab 1.5 mg Q4W | PML Safety Monitoring
Started | 0 | 0 | 0 | 13
Completed | 0 | 0 | 0 | 4
Not Completed | 0 | 0 | 0 | 9
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Etrolizumab Q4W: Etrolizumab 1.5 mg/kg was administered by SC injection Q4W for a total of 4 doses over the course of the 24-week randomized treatment phase (16-week treatment plus 8-week safety follow-up).
- Etrolizumab Q8W: Etrolizumab 3.0 mg/kg was administered by SC injection Q8W for a total of 2 doses over the course of the 24-week randomized treatment phase (16-week treatment plus 8-week safety follow-up).
- Total: Total of all reporting groups
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.25 (3.62) | 13.42 (4.46) | 12.83 (4.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 12 | 24
Disease Indication: Crohn's Disease or Ulcerative Colitis [Count of Participants; unit: Participants]
  Crohn's Disease | 5 | 5 | 10
  Ulcerative Colitis | 7 | 7 | 14
Randomization Stratification Factor: Body Weight <40 kg or ≥40 kg [Count of Participants; unit: Participants]
  <40 kg | 5 | 4 | 9
  ≥40 kg | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration (Cmax) of Etrolizumab After First and Last Dose During the Randomized Treatment Phase
Description: Etrolizumab concentrations in all pharmacokinetics (PK) samples were measured using a validated assay method. Non-compartmental analysis methods were employed to calculate PK parameters.
Time Frame: Arm Etro Q4W: Day 1, 84 and Arm Etro Q8W: Day 1, 56
Population: Pharmacokinetics (PK) Evaluable Population: all participants who received at least one dose of study drug and had evaluable PK data. This analysis included data from participants who had received their first dose (Day 1 for both arms) and last dose (on Day 56 for Q8W arm and Day 84 for Q4W arm) of study drug.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (μg/mL)
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W
Number analyzed (Participants) | 11 | 12
micrograms per millilitre (μg/mL)
  After First Dose (Day 1): number analyzed (Participants) | 10 | 12
  After First Dose (Day 1) | 7.73 (2.18) | 19.0 (8.21)
  After Last Dose (Q4W Day 84, Q8WDay 56): number analyzed (Participants) | 11 | 11
  After Last Dose (Q4W Day 84, Q8WDay 56) | 9.80 (4.86) | 18.1 (6.25)

2. Primary Outcome: Time to Maximum Serum Concentration (Tmax) of Etrolizumab After First and Last Dose During the Randomized Treatment Phase
Description: as for outcome 1
Time Frame: Arm Etro Q4W: Days 1, 84 and Arm Etro Q8W: Days 1, 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W
Number analyzed (Participants) | 11 | 12
Day
  After First Dose (Day 1): number analyzed (Participants) | 10 | 12
  After First Dose (Day 1) | 4.65 (1.43) | 4.00 (1.48)
  After Last Dose (Q4W Day 84, Q8WDay 56): number analyzed (Participants) | 11 | 11
  After Last Dose (Q4W Day 84, Q8WDay 56) | 5.04 (2.92) | 4.94 (3.28)

3. Primary Outcome: Area Under the Concentration-Time Curve Within the Last Dosing Interval (AUC-tau) of Etrolizumab During the Randomized Treatment Phase
Description: as for outcome 1
Time Frame: Arm Etro Q4W: Days 56, 84, 88, 98, 112 and Arm Etro Q8W: Day 56, 60, 70, 84, 88, 98, 112
Population: Pharmacokinetics (PK) Evaluable Population: all participants who received at least one dose of study drug and had evaluable PK data. This analysis included data from participants who had received their last dose of study drug (on Day 56 for Q8W arm and Day 84 for Q4W arm).
Measure: Mean (Standard Deviation); unit: Day*μg/mL
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W
Number analyzed (Participants) | 11 | 12
Day*μg/mL
  AUC56-112: number analyzed (Participants) | 0 | 10
  AUC56-112 |  | 521 (306)
  AUC84-112: number analyzed (Participants) | 11 | 0
  AUC84-112 | 167 (86.9) |

4. Primary Outcome: Elimination Half-Life (t1/2) of Etrolizumab After Last Dose During the Randomized Treatment Phase
Description: as for outcome 1
Time Frame: Arm Etro Q4W: Days 84, 88, 98, 112, 126, 140, 168 and Arm Etro Q8W: Days 56, 60, 70, 84, 88, 98, 112, 126, 140, 168
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W
Number analyzed (Participants) | 11 | 10
Day | 7.31 (1.76) | 8.65 (3.74)

5. Primary Outcome: Serum Trough Concentration (Ctrough) of Etrolizumab at the End of Each Dosing Interval During the Randomized Treatment Phase
Description: Etrolizumab concentrations in all pharmacokinetics (PK) samples were measured using a validated assay method.
Time Frame: Arm Etro Q4W: Predose on Days 28, 56, 84, 112 and Arm Etro Q8W: Predose on Days 56, 112
Population: Pharmacokinetics (PK) Evaluable Population: all participants who received at least one dose of study drug and had evaluable PK data. This analysis included data from participants at the end of each dosing interval (on Days 28, 56, 84, and 112 for Q4W arm and Days 56 and 112 for Q8W arm).
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (μg/mL)
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W
Number analyzed (Participants) | 11 | 12
micrograms per millilitre (μg/mL)
  Day 28: number analyzed (Participants) | 11 | 0
  Day 28 | 1.87 (1.32) |
  Day 56: number analyzed (Participants) | 11 | 11
  Day 56 | 3.22 (2.24) | 1.82 (1.99)
  Day 84: number analyzed (Participants) | 11 | 0
  Day 84 | 3.00 (2.38) |
  Day 112: number analyzed (Participants) | 11 | 10
  Day 112 | 2.79 (2.01) | 3.70 (4.64)

6. Primary Outcome: Percentage of Baseline Absolute Numbers of Beta7 Receptor-Expressing Gut Homing CD3, CD4, and CD8 T Cells and CD19 B Cells With Unoccupied Beta7 Receptors in Peripheral Blood, Assessed by Flow Cytometry, During the Randomized Treatment Phase
Description: Target engagement of etrolizumab was assessed via measurement of Beta7 receptor occupancy on Beta7 receptor-expressing gut homing lymphocyte subsets in peripheral blood, including CD3, CD4, and CD8 T cells and CD19 B cells, using qualified flow cytometry methods. A decrease to 0% of baseline (BL) in median absolute cell counts of Beta7 receptor-expressing T and B cell subsets with unoccupied Beta7 receptors following etrolizumab treatment indicated maximal receptor occupancy by etrolizumab.
Time Frame: Predose (dosing days only) at Baseline (Day 1) and on Days 4, 56, 84, 98, and 112 (Treatment Period), and Days 126, 140, and 168 (Follow-Up Period)
Population: Pharmacodynamics (PD) Evaluable Population: all participants who received at least one dose of study treatment and had evaluable PD data.
Measure: Median (Standard Deviation); unit: Percentage of BL Unoccupied Beta7 Cells
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W
Number analyzed (Participants) | 12 | 12
Percentage of BL Unoccupied Beta7 Cells
  CD3 T Cells: Baseline: number analyzed (Participants) | 11 | 10
  CD3 T Cells: Baseline | 100 (0.0) | 100 (0.0)
  CD3 T Cells: Day 4: number analyzed (Participants) | 8 | 10
  CD3 T Cells: Day 4 | 0.18 (0.2) | 0.40 (0.4)
  CD3 T Cells: Day 56: number analyzed (Participants) | 9 | 10
  CD3 T Cells: Day 56 | 1.92 (1.9) | 13.74 (13.5)
  CD3 T Cells: Day 84: number analyzed (Participants) | 9 | 9
  CD3 T Cells: Day 84 | 7.43 (6.0) | 1.06 (1.1)
  CD3 T Cells: Day 98: number analyzed (Participants) | 10 | 9
  CD3 T Cells: Day 98 | 0.36 (0.4) | 1.06 (1.1)
  CD3 T Cells: Day 112: number analyzed (Participants) | 10 | 9
  CD3 T Cells: Day 112 | 4.06 (2.6) | 6.01 (5.6)
  CD3 T Cells: Day 126: number analyzed (Participants) | 9 | 8
  CD3 T Cells: Day 126 | 12.00 (12.0) | 27.24 (24.6)
  CD3 T Cells: Day 140: number analyzed (Participants) | 9 | 9
  CD3 T Cells: Day 140 | 47.47 (21.9) | 56.82 (22.2)
  CD3 T Cells: Day 168: number analyzed (Participants) | 10 | 9
  CD3 T Cells: Day 168 | 71.64 (22.4) | 51.79 (23.1)
  CD4 T Cells: Baseline: number analyzed (Participants) | 11 | 10
  CD4 T Cells: Baseline | 100 (0.0) | 100 (0.0)
  CD4 T Cells: Day 4: number analyzed (Participants) | 8 | 10
  CD4 T Cells: Day 4 | 0.17 (0.2) | 0.00 (0.0)
  CD4 T Cells: Day 56: number analyzed (Participants) | 9 | 10
  CD4 T Cells: Day 56 | 3.33 (3.3) | 16.56 (16.1)
  CD4 T Cells: Day 84: number analyzed (Participants) | 9 | 9
  CD4 T Cells: Day 84 | 7.14 (7.1) | 1.28 (1.0)
  CD4 T Cells: Day 98: number analyzed (Participants) | 10 | 9
  CD4 T Cells: Day 98 | 0.24 (0.2) | 1.28 (1.3)
  CD4 T Cells: Day 112: number analyzed (Participants) | 10 | 9
  CD4 T Cells: Day 112 | 3.60 (3.1) | 6.74 (6.4)
  CD4 T Cells: Day 126: number analyzed (Participants) | 9 | 8
  CD4 T Cells: Day 126 | 13.33 (13.3) | 37.03 (33.7)
  CD4 T Cells: Day 140: number analyzed (Participants) | 9 | 9
  CD4 T Cells: Day 140 | 55.34 (23.9) | 62.01 (20.3)
  CD4 T Cells: Day 168: number analyzed (Participants) | 10 | 9
  CD4 T Cells: Day 168 | 74.49 (26.1) | 50.00 (16.3)
  CD8 T Cells: Baseline: number analyzed (Participants) | 11 | 10
  CD8 T Cells: Baseline | 100 (0.0) | 100 (0.0)
  CD8 T Cells: Day 4: number analyzed (Participants) | 8 | 10
  CD8 T Cells: Day 4 | 0.00 (0.0) | 0.00 (0.0)
  CD8 T Cells: Day 56: number analyzed (Participants) | 9 | 10
  CD8 T Cells: Day 56 | 1.56 (1.6) | 8.41 (8.4)
  CD8 T Cells: Day 84: number analyzed (Participants) | 9 | 9
  CD8 T Cells: Day 84 | 2.72 (2.7) | 0.00 (0.0)
  CD8 T Cells: Day 98: number analyzed (Participants) | 10 | 9
  CD8 T Cells: Day 98 | 1.10 (1.1) | 2.33 (2.3)
  CD8 T Cells: Day 112: number analyzed (Participants) | 10 | 9
  CD8 T Cells: Day 112 | 0.97 (1.0) | 2.46 (2.5)
  CD8 T Cells: Day 126: number analyzed (Participants) | 9 | 8
  CD8 T Cells: Day 126 | 20.00 (20.0) | 14.51 (14.5)
  CD8 T Cells: Day 140: number analyzed (Participants) | 9 | 9
  CD8 T Cells: Day 140 | 54.17 (18.8) | 40.98 (24.7)
  CD8 T Cells: Day 168: number analyzed (Participants) | 10 | 9
  CD8 T Cells: Day 168 | 63.34 (40.1) | 55.56 (21.1)
  CD19 B Cells: Baseline: number analyzed (Participants) | 11 | 10
  CD19 B Cells: Baseline | 100 (0.0) | 100 (0.0)
  CD19 B Cells: Day 4: number analyzed (Participants) | 8 | 10
  CD19 B Cells: Day 4 | 0.00 (0.0) | 0.00 (0.0)
  CD19 B Cells: Day 56: number analyzed (Participants) | 9 | 10
  CD19 B Cells: Day 56 | 3.57 (3.6) | 19.14 (17.1)
  CD19 B Cells: Day 84: number analyzed (Participants) | 9 | 9
  CD19 B Cells: Day 84 | 10.71 (10.7) | 0.00 (0.0)
  CD19 B Cells: Day 98: number analyzed (Participants) | 10 | 9
  CD19 B Cells: Day 98 | 0.00 (0.0) | 0.00 (0.0)
  CD19 B Cells: Day 112: number analyzed (Participants) | 9 | 9
  CD19 B Cells: Day 112 | 7.14 (7.1) | 7.14 (7.1)
  CD19 B Cells: Day 126: number analyzed (Participants) | 9 | 8
  CD19 B Cells: Day 126 | 42.86 (21.4) | 33.93 (32.3)
  CD19 B Cells: Day 140: number analyzed (Participants) | 9 | 9
  CD19 B Cells: Day 140 | 68.00 (30.5) | 77.78 (32.6)
  CD19 B Cells: Day 168: number analyzed (Participants) | 10 | 9
  CD19 B Cells: Day 168 | 73.21 (17.7) | 40.00 (13.2)

7. Secondary Outcome: Number of Participants With Adverse Events by Highest Severity Grade, Assessed According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI-CTCAE v4.0), During the Randomized Treatment Phase
Description: All adverse events (AEs) were graded for severity using the NCI-CTCAE v4.0. Any AE not specifically listed was assessed per the following 5 grades: Grade 1 = mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated. Grade 2 = moderate; minimal, local, or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living. Grade 3 = severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living. Grade 4 = life-threatening consequences or urgent intervention indicated. Grade 5 = death related to AE. Not all grades are appropriate for all AEs; some AEs have fewer than 5 options. The terms "severe" and "serious" are not synonymous and are independently assessed for each AE. Multiple occurrences of AEs were counted only once per participant at the highest (worst) grade.
Time Frame: From Baseline until 12 weeks (Q4W arm only) or 16 weeks (Q8W arm only) after the last dose of study drug during the randomized treatment phase (up to 24 weeks)
Population: Safety Population: all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W
Number analyzed (Participants) | 12 | 12
Participants
  Any Adverse Event - Any Grade | 9 | 10
  Any Adverse Event - Grade 1 | 2 | 2
  Any Adverse Event - Grade 2 | 4 | 5
  Any Adverse Event - Grade 3 | 3 | 3
  Any Adverse Event - Grade 4 | 0 | 0
  Any Adverse Event - Grade 5 | 0 | 0

8. Secondary Outcome: Number of Participants With Serious Infection-Related Adverse Events During the Randomized Treatment Phase
Description: Serious infection-related AEs were assessed using NCI-CTCAE v4.0.
Time Frame: as for outcome 7
Population: Safety Population: all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Hypersensitivity Reactions During the Randomized Treatment Phase
Description: Hypersensitivity reactions were assessed using NCI-CTCAE v4.0.
Time Frame: as for outcome 7
Population: Safety Population: all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Malignancies During the Randomized Treatment Phase
Description: Malignancies were assessed using NCI-CTCAE v4.0.
Time Frame: as for outcome 7
Population: Safety Population: all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) to Etrolizumab at Baseline and Post-Baseline During the Randomized Treatment Phase
Description: Participants were considered to be etrolizumab anti-drug antibody (ADA) positive if they were ADA negative or had missing data at Baseline (BL) but developed an ADA response following study drug exposure (i.e., treatment-induced ADA positive), or if they were ADA positive at baseline and the titer of one or more postbaseline samples was at least 0.60 titer unit greater than the titer of the baseline sample (i.e., treatment-enhanced ADA positive); these ADA positive responses are summarized together (induced + enhanced) in the 'treatment-emergent ADA positive' category. Participants were considered to be ADA negative if they were ADA negative or had missing data at Baseline (BL) and all postbaseline samples were negative (i.e., treatment-emergent ADA negative).
Time Frame: Predose (dosing days only) on Days 1, 28, 84, 112, and 168 (up to the end of the randomized treatment phase at Week 24)
Population: ADA Evaluable Population: all participants who received at least one dose of study treatment and had at least one baseline or post-baseline ADA result from at least one sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W
Number analyzed (Participants) | 12 | 12
Participants
  Baseline (BL): ADA Positive | 1 | 0
  BL: ADA Negative | 11 | 12
  Post-BL: Treatment-Emergent ADA Positive: number analyzed (Participants) | 11 | 12
  Post-BL: Treatment-Emergent ADA Positive | 4 | 2
  Post-BL: Treatment-Emergent ADA Negative: number analyzed (Participants) | 11 | 12
  Post-BL: Treatment-Emergent ADA Negative | 7 | 10

12. Secondary Outcome: Long-Term Safety of Etrolizumab: Number of Participants With Adverse Events by Highest Severity Grade, Assessed According to NCI-CTCAE v4.0
Description: as for outcome 7
Time Frame: OLE Period: From end of Week 24 to end of 12-week safety follow-up (up to 195 weeks); PML Period: After completion of safety follow up in Randomized Treatment phase or after completion of safety follow up after OLE treatment, up to approximately 92 weeks
Population: Safety Population: all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE: Etrolizumab 1.5 mg Q4W | PML Safety Monitoring
Number analyzed (Participants) | 21 | 13
Participants
  Any Adverse Event - Any Grade | 20 | 4
  Any Adverse Event - Grade 1 | 0 | 2
  Any Adverse Event - Grade 2 | 12 | 2
  Any Adverse Event - Grade 3 | 8 | 0
  Any Adverse Event - Grade 4 | 0 | 0
  Any Adverse Event - Grade 5 | 0 | 0

13. Secondary Outcome: Long-Term Safety of Etrolizumab: Number of Participants With Serious Infection-Related Adverse Events
Description: Serious infection-related AEs were assessed using NCI-CTCAE v4.0.
Time Frame: as for outcome 12
Population: Safety Population: all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE: Etrolizumab 1.5 mg Q4W | PML Safety Monitoring
Number analyzed (Participants) | 21 | 13
Participants | 1 | 0

14. Secondary Outcome: Long-Term Safety of Etrolizumab: Number of Participants With Hypersensitivity Reactions
Description: Hypersensitivity reactions were assessed using NCI-CTCAE v4.0.
Time Frame: as for outcome 12
Population: Safety Population: all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE: Etrolizumab 1.5 mg Q4W | PML Safety Monitoring
Number analyzed (Participants) | 21 | 13
Participants | 4 | 1

15. Secondary Outcome: Long-Term Safety of Etrolizumab: Number of Participants With Malignancies
Description: Malignancies were assessed using NCI-CTCAE v4.0.
Time Frame: as for outcome 12
Population: Safety Population: all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE: Etrolizumab 1.5 mg Q4W | PML Safety Monitoring
Number analyzed (Participants) | 21 | 13
Participants | 0 | 0

16. Secondary Outcome: Long-Term Safety of Etrolizumab: Number of Participants With Anti-Drug Antibodies (ADAs) to Etrolizumab at Baseline and Post-Baseline
Description: as for outcome 11
Time Frame: Predose (dosing days only) at Baseline (Day 1), Days 28, 84, and 112, Weeks 24, 36, 72, and 120, and every 12 weeks thereafter for up to 4.25 years
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Groups:
- Etrolizumab Q4W: Etrolizumab 1.5 milligrams mg/kg was administered by SC injection Q4W for a total of 4 doses over the course of the 24-week randomized treatment phase (16-week treatment plus 8-week safety follow-up). Thereafter, participants were given the option to participate in the OLE period to receive etrolizumab 1.5 mg/kg SC Q4W for maximum of 183 weeks. After the randomized treatment period or OLE period participants who chose to enroll in the PML safety surveillance phase were monitored for PML for approximately 92 weeks.
- Etrolizumab Q8W: Etrolizumab 3.0 mg/kg was administered by SC injection once Q8W for a total of 2 doses over the course of the 24-week randomized treatment phase (16-week treatment plus 8-week safety follow-up). Thereafter, participants were given the option to participate in the week OLE period to receive etrolizumab 1.5 mg/kg SC Q4W for maximum of 183 weeks. After the randomized treatment period or OLE period participants who chose to enroll in PML safety surveillance phase were monitored for PML for approximately 92 weeks.
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W
Number analyzed (Participants) | 12 | 12
Participants
  Baseline (BL): ADA Positive | 1 | 0
  BL: ADA Negative | 11 | 12
  Post-BL: Treatment-Emergent ADA Positive: number analyzed (Participants) | 11 | 12
  Post-BL: Treatment-Emergent ADA Positive | 4 | 3
  Post-BL: Treatment-Emergent ADA Negative: number analyzed (Participants) | 11 | 12
  Post-BL: Treatment-Emergent ADA Negative | 7 | 9

17. Secondary Outcome: Number of Participants With Confirmed Progressive Multifocal Leukoencephalopathy (PML) During the Post-Treatment PML Monitoring Phase
Description: The safety surveillance PML-monitoring phase (no etrolizumab treatment) consisted of telephone calls approximately every 6 months with administration of the protocol's PML Subjective Checklist. If there were any signs or symptoms suggestive of PML identified on this subjective checklist during the telephone call, the participant was asked to come into the clinic for a neurologic examination. The protocol's PML Algorithm was followed for any suspected case of PML, and any confirmed case of PML would be reported as a serious adverse event.
Time Frame: PML Period: After completion of safety follow up in Randomized Treatment period or after completion of safety follow up after OLE treatment, up to approximately 92 weeks
Population: Safety Population: all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PML Safety Monitoring
Number analyzed (Participants) | 13
Participants | 0

ADVERSE EVENTS:
Time Frame: From Baseline up to the last dose of drug in the Randomized Treatment phase (up to 24 weeks); OLE Period: From end of Week 24 up to end of 12-week safety follow-up (up to 195 weeks); PML Period: After completion of safety follow up in the Randomized Treatment phase or after completion of safety follow up after OLE treatment, up to approximately 92 weeks
Description: After informed consent but prior to initiation of study drug, only serious AEs caused by protocol-mandated intervention were reported. After initiation of study drug, all AEs were reported until the last study visit or 12 weeks after the last dose of study drug. After this period, only serious AEs related to prior study drug were reported. Safety population included all treated participants in the study.
Groups:
- OLE: Etrolizumab 1.5 mg/kg Q4W: Participants from Etrolizumab Q4W and Etrolizumab Q8W who completed the randomized treatment period, were given the option to participate in the OLE period. All participants who chose to enter the OLE period were administered etrolizumab 1.5 mg/kg SC Q4W for a maximum of 183 weeks. Post treatment discontinuation patients entered a 12-week safety follow up.
Arm/Group | Etrolizumab Q4W | Etrolizumab Q8W | OLE: Etrolizumab 1.5 mg/kg Q4W | PML Safety Monitoring
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/21 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/12 | 2/12 | 6/21 | 0/13
Other Adverse Events (participants affected / at risk) | 8/12 | 9/12 | 20/21 | 4/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etrolizumab Q4W (N=12) | Etrolizumab Q8W (N=12) | OLE: Etrolizumab 1.5 mg/kg Q4W (N=21) | PML Safety Monitoring (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Idiopathic intracranial hypertension (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etrolizumab Q4W (N=12) | Etrolizumab Q8W (N=12) | OLE: Etrolizumab 1.5 mg/kg Q4W (N=21) | PML Safety Monitoring (N=13)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 4 (5) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (4) | 6 (12) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (5) | 2 (2)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (3) | 2 (3) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2) | 0 (0) | 7 (13) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 2 (2) | 2 (2) | 5 (9) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (7) | 0 (0) | 6 (6) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (3) | 2 (5) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (7) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 8 (16) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 2 (2) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (4) | 5 (8) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Polymenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vaccination site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT03478956/Prot_SAP_001.pdf